CLINICAL TRIAL: NCT06121245
Title: Evaluating the Release of the Entero-pancreatic Hormone Somatostatin by Measuring Stable Co-secreted Prosomatostatin Moieties in the Plasma of Healthy Individuals - the PRO-SOma COla (PROSOCO) Study
Brief Title: The PRO-SOma COla (PROSOCO) Study
Acronym: PROSOCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Simon Veedfald, Assistant professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PROSOCO
Record Dates: First submitted 2023-10-18; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: somatostatin; secretion; peptide; pro-somatostatin 1-64
MeSH Terms: interventions — Proton Pump Inhibitors

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, crossover study
Who Masked: Participant, Investigator
Masking Description: Pharmacy prepared placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esomeprazol (Experimental): On the day before the study visits participants will ingest a capsule in the morning on a capsule in the evening containing Esomperazol
  Interventions: Other: Proton Pump inhibitor
- Placebo (Placebo Comparator): On the day before the study visits participants will ingest a capsule in the morning on a capsule in the evening containing a placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Proton Pump inhibitor — A proton pump inhibitor will be used as a tool to study the effect of pH changes in the stomach lumen on the release of somatostatin (evaluated by measurements of somatostatin and pro-somatostatin 1-64)
  Arms: Esomeprazol
Other: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled, crossover study is to determine whether it is possible to gauge the pattern of somatostatin secretion by measuring plasma concentrations of pro-somatostatin 1-64 (a stable peptide that is released in equimolar amounts alongside somatostatin) as a surrogate marker. During the study the release of somatostatin will be manipulated by changing the luminal pH of the stomach.

Healthy participants will be studied in a randomized on two occasions. The day before both two study visits participants will ingest a capsule in the morning and a capsule in the evening. On one day the capsule will contain a proton pump inhibitor (Esomeprazol) to elevate the luminal pH of the stomach and on the other day the capsule will be a placebo. On the study days participants will ingest, in the mornng after an overnight fast, a coca cola zero + lemon juice to lower the luminal pH which willelicit the release of somatostatin. Blood samples will be collected before and after the ingestion of coca cola.

DETAILED DESCRIPTION:
Somatostatin is a polypeptide that plays a key regulatory role in the gastrointestinal tract and pancreas. It has been attempted to determine in peripheral plasma samples the pattern of somatostatin release. However, due to the brief half-life of somatostatin this it turns out is difficult. Therefore, the investigators have developed an antibodies and a radioimmunoassay that measures concentrations of a stable peptide termed prosomatostatin 1-64. This peptide is released in equimolar amounts alongside somatostatin from the somatostatin-producing cells in the gut.

The current study aims to demonstrate that prosomatostatin 1-64 can be picked up in peripheral plasma from human study participants. The release of somatostatin is increased when the pH of the stomach is low. The release of somatostatin will be elicited by asking participants coca cola zero with lemon juice. Participants will be studied on two occasions (on one day participants will be pretreated with a proton pump inhibitor, on the other day with a placebo). The two visits will be carried out as a placebo-controlled crossover study following a randomised schedule.

If successful, pro-somatostatin 1-64 can be as a surrogate marker of somatostatin secretion. This will allow investigations of somatostatin secretion dynamics in humans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Non-diabetic fasting plasma glucose (< 7.0 mmol/L) at time of inclusion
* Normal weight and weight stable
* Written informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Haemoglobin < 7.9 mmol/L
* Prior gastrointestinal operations excluding uncomplicated appendectomy
* Significant gastrointestinal symptoms (e.g. dyspepsia, postprandial pain)
* Intolerance to aspartame
* Use of medication that may influence blood pressure, gastrointestinal motor function, body weight or appetite (e.g. antihypertensive drugs, anticholinergic drugs (e.g. atropine, hyoscine), prokinetic drugs (metoclopramide, domperidone, erythromycin), orlistat, green tea extracts, astragalus, St. John's Wort etc.)
* Evidence of drug abuse, consumption of tobacco in any form or daily consumption of more than 20g alcohol
* History of gastrointestinal disease, including significant upper or lower gastrointestinal symptoms, pancreatitis, or previous gastrointestinal surgery including cholecystectomy (but not uncomplicated appendectomy) Participation in any other research studies within the previous 3 months
* Inability to give informed consent
* Non-Probability Sample: Any of a variety of other sampling processes, such as convenience sampling or invitation to volunteer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of pro-somatostatin 1-64 | baseline samples, 7, 10, 15, 20, 25, 30, 45, 60, 90, 120 min
  Peptide released from D-cells in the gut in equimolar concentrations alongside somatostatin

SECONDARY OUTCOMES:
Plasma concentration of gastrin | baseline samples, 7, 10, 15, 20, 25, 30, 45, 60, 90, 120 min
  peptide hormone released from G cells in the antrum of the stomach
Plasma concentration of cholecystokinin | baseline samples, 7, 10, 15, 20, 25, 30, 45, 60, 90, 120 min
  peptide hormone released from I cells in the proximal small intestine
Plasma concentration of secretin | baseline samples, 7, 10, 15, 20, 25, 30, 45, 60, 90, 120 min
  Peptide hormone released from S cells in the small intestine
Plasma concentration of pancreatic polypeptide | baseline samples, 7, 10, 15, 20, 25, 30, 45, 60, 90, 120 min
  Peptide hormone released from the endocrine pancreas
Plasma concentration of glucose | baseline samples, 7, 10, 15, 20, 25, 30, 45, 60, 90, 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Jens J Holst, MD, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - University of Copenhagen, Copenhagen, Capital
  - Hvidovre University Hospital, Hvidovre, Capital